CLINICAL TRIAL: NCT00904787
Title: A Phase 1 Study of ENMD-2076 in Patients With Relapsed or Refractory Hematological Malignancies
Brief Title: Study of ENMD-2076 in Patients With Relapsed or Refractory Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Carolyn Sidor, Chief Medical Officer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2076-CL-003
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Relapsed or Refractory Hematological Malignancies
Keywords: Leukemia; Hematologic neoplasms
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms; Leukemia | interventions — ENMD 2076

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076 — capsule, dose escalation, taken orally, daily in 28 day cycles

SUMMARY:
To define the maximum tolerated dose of oral daily ENMD 2076 in patients with relapsed or refractory hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed/refractory hematological malignancy for which no standard therapies are anticipated to result in a durable remission. Patients with poor-risk myelodysplasia (MDS) [i.e., IPSS ≥ 1.5] or chronic myelomonocytic leukemia (CMML) are also candidates for this protocol. Relapsed/refractory leukemias include acute non lymphocytic leukemia (AML) by WHO classification, acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blast crisis. Patients with agnogenic myeloid metaplasia (AMM) are also eligible. Patients with relapsed or refractory lymphoma or myeloma may also participate.
* Age ≥18 years.
* Adequate performance status
* Interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents and adequate recovery from prior toxicities. If the patient had a transplant, at least 6 months must have passed before initiation of treatment on this protocol and stable graft versus host disease (no change in severity) for 4 weeks preceding study entry (if applicable).
* Persistent clinically significant chronic toxicities from prior therapy must have resolved to baseline or NCI CTCAE Grade < 1
* Adequate laboratory results within 10 days of ENMD-2076 administration (unless the abnormality is considered attributable to leukemia)

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Clinical evidence of bowel obstruction, active uncontrolled malabsorption syndromes or a history of total gastrectomy.
* Impaired cardiac function including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, uncontrolled hypertension, or uncontrolled congestive heart failure. Blood pressure must be < 150/90 at the time of enrollment.
* Receiving any other treatment for their disease
* QTc prolongation defined as ≥ 470 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Define the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of oral daily ENMD 2076 by evaluation of adverse events | Day 1 through first cycle of therapy

SECONDARY OUTCOMES:
Safety and toxicity of repeated oral dosing of ENMD 2076 | Throughout study participation
Describe any preliminary evidence of anti-cancer effects of ENMD-2076 in patients with hematological malignancies | monthly

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada